CLINICAL TRIAL: NCT02471274
Title: A Phase 1, Open-label, Parallel-group Study to Evaluate the Single-dose Pharmacokinetics of Sotagliflozin in Male and Female Subjects With Mild, Moderate, and Severe Hepatic Impairment and Matched Subjects With Normal Hepatic Function
Brief Title: PK Study of Sotagliflozin in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-116-HEP; LX4211.116 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): healthy control subjects with normal hepatic function
  Interventions: Drug: sotagliflozin
- Group 2 (Experimental): subjects with mild hepatic impairment
  Interventions: Drug: sotagliflozin
- Group 3 (Experimental): subjects with moderate hepatic impairment
  Interventions: Drug: sotagliflozin
- Group 4 (Experimental): subjects with severe hepatic impairment
  Interventions: Drug: sotagliflozin

INTERVENTIONS:
Drug: sotagliflozin — single 400 mg dose

SUMMARY:
To evaluate the effect of mild, moderate, or severe hepatic impairment on the pharmacokinetics (PK) of a single dose of 400 mg sotagliflozin (2 x 200-mg tablets) compared with healthy, demographically-matched subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects ≥18 to ≤70 years of age
* Body mass index ≥18.0 to ≤36.0 kg/m2, inclusive, at Screening
* Subjects with mild, moderate, or severe hepatic impairment
* Control group of matched healthy subjects
* Willing and able to provide written informed consent

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or ECG findings that may interfere with any aspect of study conduct or interpretation of results
* Existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism, or excretion of sotagliflozin
* History of any major surgery within 6 months
* History of renal disease, or significantly abnormal kidney function test
* Women who are breastfeeding or are planning to become pregnant during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of sotaglifozin to evaluate protocol specified PK parameters | Day 1 to Day 5

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | Day 1 to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Lexicon Investigational Site, Lakewood, Colorado
  - Lexicon Investigational Site, Miami, Florida
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, Minneapolis, Minnesota